CLINICAL TRIAL: NCT06849180
Title: Novel Subtypes and Treatment Strategies of Patients with Unresectable Mixed Hepatocellular Cholangiocarcinoma Based on Multimodal Data
Brief Title: Novel Subtypes and Treatment Strategies of Patients with Unresectable Combined Hepatocellular Cholangiocarcinoma Based on Multimodal Data
Status: Recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Jiangsu Cancer Institute & Hospital (Other); Yunnan Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Shanghai Zhongshan Hospital (Other); Sun Yet-Sen University Cancer Center (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of interventional and Vascular Surgery Department, Zhongda Hospital
Other Study IDs: 2024040195
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Combined Hepatocellular-cholangiocarcinoma; Combined Hepatocellular Carcinoma and Cholangiocarcinoma; Combined Hepatocellular and Cholangiocarcinoma
Keywords: CHC; cHCC-ICC
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Combination Product: Interventional therapies combined with or without systemic drugs — The study will include adult patients with histologically/cytologically confirmed unresectable CHC. Collect patient genomics, proteomics, immune microenvironment, pathology reports, medical images and clinical electronic medical records, etc., to form high-quality and deeply labeled data sets to support the subsequent development and application of AI large models. Based on multi-source heterogeneous data of CHC patients, a large model for comprehensive diagnosis and treatment was constructed. Firstly, multi-modal data of different stages of disease were integrated by using cross-modal multi-course fusion technology to achieve efficient fusion of complex data. Secondly, by fine-tuning the large model, tasks such as CHC classification, prognosis inference and treatment plan recommendation are accurately completed, and potential information in the diagnosis and treatment process is mined.

SUMMARY:
This study focused on exploring new comprehensive treatment strategies for patients with unresectable combined hepatocellular-cholangiocarcinoma, classifying patients with CHC subtypes based on the combination of artificial intelligence and multi-omics, and exploring the optimal treatment strategies for patients with different subtypes, helping clinicians to screen the most beneficial groups of various treatment schemes, and providing new ideas for safe treatment of high-risk patients.

DETAILED DESCRIPTION:
This will be a multicenter observational study that will be conducted at several leading liver cancer treatment centers. The study will include adult patients with histologically/cytologically confirmed unresectable CHC. Collect patient genomics, proteomics, immune microenvironment, pathology reports, medical images and clinical electronic medical records, etc., to form high-quality and deeply labeled data sets to support the subsequent development and application of AI large models. Based on multi-source heterogeneous data of CHC patients, a large model for comprehensive diagnosis and treatment was constructed. Firstly, multi-modal data of different stages of disease were integrated by using cross-modal multi-course fusion technology to achieve efficient fusion of complex data. Secondly, by fine-tuning the large model, tasks such as CHC classification, prognosis inference and treatment plan recommendation are accurately completed, and potential information in the diagnosis and treatment process is mined.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years; diagnosis of CHC confirmed by histology or cytology;
2. patients with unresectable or metastatic CHC diagnosed on the basis of unresectable CHC who have received prior local therapy, systemic therapy, or a combination of both and have at least one measurable lesion (RECIST v1.1);
3. survival time ≥ 3 months;
4. ECOG PS 0-2;
5. Child-Pugh A/B.

Exclusion Criteria:

1. pregnant women, lactating women, and men and women of childbearing age who are unwilling or unable to use effective contraception.
2. history of other malignant tumors within the past five years, unless these tumors have been completely treated and have been free of active disease for five years prior to the first dose and are at low risk of recurrence.
3. fully treated carcinoma in situ with no evidence of disease.
4. history of gastrointestinal bleeding or significant bleeding tendency (e.g., with known active ulcers, fecal occult blood, etc.) within the past six months that precludes inclusion in the study; gastroscopy is required if there is persistent fecal occult blood.
5. substantial organ transplantation or bone marrow transplantation within two years prior to the first dose, or active autoimmune disease requiring systemic therapy.
6. other conditions that the investigator deems unsuitable for inclusion in the study. Inadequate information, such as incomplete data from laboratory tests, missing or poor quality imaging data, no prognostic information, etc., that the investigator considers unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for the planned retrospective analysis of this project is patients with pathologically confirmed mixed hepatocellular cholangiocarcinoma, based on the 2024 NCCN Clinical Practice Guidelines in Oncology: Hepatocellular Carcinoma [Version 2.2024]) and China's Primary Liver Cancer Diagnosis and Treatment Guidelines (2024) are defined as unresectable patients.
Sampling Method: Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to RECIST 1.1) or death due to any cause, whichever occurs first.
PFS per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Objective response rate(ORR) per RESCIST 1.1 | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR per mRECIST | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
Duration of Response (DOR) per RESCIST 1.1 | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to RESCIST 1.1) or death due to any cause, whichever occurs first.
DOR per mRECIST | up to approximately 2 years
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR or PR until the first documented disease progression (according to mRECIST) or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) per RESCIST 1.1 | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD)per RESCIST 1.1.
DCR per mRECIST | up to approximately 2 years
  DCR is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD) per mRECIST.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China